CLINICAL TRIAL: NCT06735820
Title: Early Phase Study to Evaluate the MEK Inhibitor Selumetinib With the MDM2 Inhibitor APG-115 in Patients With Neurofibromatosis Type 1 and Pre-malignant and Malignant Peripheral Nerve Sheath Tumors
Brief Title: Early Phase Study Evaluating MEK and MDM2 Inhibition in Patients With NF1 and MPNST
Acronym: MEKMDM2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AeRang Kim (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, AeRang Kim, Pediatric Oncologist, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001200; W81XWH-22-1-1120 (Other Grant/Funding Number: U.S. Army Medical Research and Development Command)
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Malignant Peripheral Nerve Sheath Tumor (MPNST); Neurofibromatosis 1 (NF1); Atypical Neurofibroma
Keywords: NF1; MPNST; MEK inhibitor; MDM2 inhibitor; atypical neurofibroma; ANNUBP
MeSH Terms: conditions — Neurofibrosarcoma; Neurofibromatosis 1 | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- APG-115 and Selumetinib (Experimental): There is only one arm. It is combination therapy of APG-115 and Selumetinib.
  Interventions: Drug: APG-115; Drug: Selumetinib

INTERVENTIONS:
Drug: APG-115 — Combination therapy of APG-115 and Selumetinib
  Other Names: alrizomadlin
Drug: Selumetinib — Combination therapy of APG-115 and Selumetinib
  Other Names: koselugo

SUMMARY:
This is a phase 0/1/2, multi-site study to evaluate the MEK inhibitor Selumetinib with the MDM2 Inhibitor APG-115 in patients with Neurofibromatosis Type 1 and pre-malignant and malignant peripheral nerve sheath tumors

DETAILED DESCRIPTION:
The first primary objective of the study is to determine the safety, tolerability, pharmacokinetics, and recommended doses of selumetinib and APG-115 in patients with Neurofibromatosis Type 1 (NF1) and refractory/unresectable MPNST (Part A). The second primary objective is to determine the clinical benefit of selumetinib and APG-115 in patients with NF1 and refractory/unresectable MPNST (Part B). The secondary objective is to evaluate the percent apoptosis and tumor proliferation in resectable atypical neurofibromatus neoplasm of uncertain biologic potential (ANNUBP) after exposure to selumetinib and APG-115 (Part C)

ELIGIBILITY:
Inclusion Criteria:

* AGE: Part A and C: ≥ 18 years of age AGE: Part B: ≥12 years (minimum BSA ≥0.55m2)
* Part A and B: Patients with unresectable or metastatic histologically confirmed NF1 associated MPNST. Part C: Patients with NF1 and ANNUBP. Diagnostic criteria based on Miettinen et al, Human Pathol:
* MEASURABLE DISEASE: Patients must have measurable disease by RECISTv1.1. Baseline radiologic scans must be performed within 4 weeks of starting treatment.
* Therapeutic options: Parts A and B: Patients must have experienced progression after one or more prior regimens of cytotoxic chemotherapy. Patients who have refused cytotoxic chemotherapy or for whom treatment on this protocol prior to receiving cytotoxic chemotherapy is felt to be in the best interest for the patient by the local investigator will also be eligible. Part C: Patients with ANNUBP that are planned for surgical resection
* PRIOR THERAPY

  * Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering on this study excluding chronic grade 1 toxicities and alopecia.
  * No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study entry.
  * Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks (≥21 days) prior to study entry (42 days if prior nitrosourea).
  * Immunotherapy: The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 4 weeks prior to study entry.
  * Anti-cancer agents not known to be myelosuppressive (e.g not associated with reduced platelets or ANC count): ≥7 days after the last dose of the agent .
  * Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.
  * Stem Cell Transplantation. At least 2 months post-autologous stem cell transplant or at least 3 months post-allogeneic transplant and recovered from toxicities without evidence of graft versus host disease and on stable doses of immunosuppressive medications, if required.
  * Growth Factors. The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be at least 2 weeks prior to study entry.
* Concurrent therapies: No other anti-cancer therapy (chemotherapy, biological therapy, radiation therapy) permitted.
* PERFORMANCE STATUS

  * Lansky/Karnofsky performance level ≥ 50% . Participants who are wheelchair bound or have limited mobility secondary to a need for mechanical breathing support (such as an airway PN requiring tracheostomy or continuous positive airway pressure) who must have a Lansky performance of ≥ 40 (Appendix related to performance status scale).
  * For patients ≥18: Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
  * Patients who are unable to walk because of paralysis or motor weakness, but who are able to use a wheelchair will be considered ambulatory for the purpose of calculating the performance score.
* HEMATOLOGIC FUNCTION

  * Hemoglobin ≥9.0 g/dL (transfusion permissible)
  * Peripheral absolute neutrophil count (ANC) of ≥1000/μL
  * Platelet count ≥75,000/μL (transfusion independent (no transfusion within at least 7 days prior to enrollment))
* HEPATIC FUNCTION

  * Total bilirubin must be ≤ 1.5 times the upper limit of normal (ULN) or ≤3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia).
  * SGOT (AST)/SGPT (ALT) must be ≤ 3.0 times ULN
* RENAL FUNCTION: Serum creatinine ≤ 1.5 times ULN or creatinine clearance >60 ml/min/1.73m2
* CARDIAC FUNCTION:

  * Normal ejection fraction by ECHO by institutional normal (within 4 weeks of enrollment)
  * QTc ≤ 450msec (within 4 weeks of enrollment)
* Fertile men and women of childbearing potential must agree to use an effective method of birth control.
* CNS DISEASE: Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of CNS metastatic disease and are without evidence of clinical progression or stable disease at 4 weeks.

Exclusion Criteria:

* History of another primary malignancy except for:

  * A malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of the study intervention and of low potential risk of recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Stable optic pathway glioma or low-grade glioma not receiving active therapy
* History of leptomeningeal carcinomatosis
* Patients receiving other anti-cancer agents are not eligible.
* Patients who cannot swallow whole pills.
* Current or prior use of immunosuppressive medications within 14 days prior to study entry. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids or local steroid injection (e.g., intra-articular injection)
* Systemic corticosteroids used at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Any recent major surgery within a minimum of 4 weeks prior to starting drug therapy. Placement of vascular access device, percutaneous tumor biopsy, or bone marrows are not considered major surgical procedures and no minimum time frame prior to starting study drug therapy is required.
* Patients who have any known severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Severely impaired lung function defined as spirometry and DLCO that is 50% of the normal predicted value corrected for hemoglobin and alveolar volume and/or O2 saturation that is 88% or less at rest on room air. For patients who do NOT have respiratory symptoms (e.g., dyspnea at rest, known requirement for supplemental oxygen), pulmonary function test is not required.
* Cardiac conditions as follows:
* Uncontrolled hypertension (blood pressure ≥≥140/90 mmHg despite medical therapy.
* For pediatric patients: blood pressure ≥95th percentile for age, height, and gender measured as described in Appendix VIII
* Known inherited coronary disease;
* For studies with pediatric patients: History of angina or acute coronary syndrome; Acute coronary syndrome within 6 months prior to starting drug therapy
* Uncontrolled angina despite medical therapy (Canadian Cardiovascular Society grade II-IV despite medical therapy (Appendix IV))
* Symptomatic heart failure NYHA Class II-IV prior or current cardiomyopathy or severe valvular disease (Appendix V)
* Prior or current cardiomyopathy including but not limited to the following

  * Known hypertrophic cardiomyopathy
  * Known arrhythmogenic right ventricular cardiomyopathy
  * Previous moderate or severe impairment of left ventricular systolic function (LVEF <45% on echocardiography or equivalent of MUGA) even if full recovery has occurred
* Symptomatic or uncontrolled atrial fibrillation despite treatment or asymptomatic sustained ventricular tachycardia.
* Active primary immunodeficiency
* Ophthalmological conditions as follows (ophthalmology exam within 4 weeks of study enrollment)
* Current or past history of retinal pigment epithelial detachment/central serous retinopathy or retinal vein occlusion
* Known intraocular pressure (IOP)>21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma.
* Any other significant abnormality on ophthalmic examination that would make the subject unsuitable for enrolment into the study, as assessed by the investigator.
* Subjects with ophthalmological findings secondary to long standing optic pathway glioma (such as visual loss, optic nerve pallor, or strabismus) or long standing orbito-temporal PN (such as vision loss, strabismus) will not be considered a significant abnormality for purposes of this study.
* Any Supplementation with vitamin E in the 7 days prior to initiation of selumetinib.
* Hypersensitivity to investigational products, or drugs with similar chemical structures to investigational products.
* Patients unwilling or unable to comply with the protocol.
* Seville orange, star fruit, grapefruit juice, St. Johns' Wort use are not allowed while on study.
* Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of selumetinib.
* Receiving herbal supplements or medications known to be strong or moderate inhibitors or inducers of the cytochrome P450 (CYP)2C19 and CYP3A4 enzymes or fluconazole unless such products can be safely discontinued at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication.
* Persistent toxicities (CTCAE Grade ≥2) caused by previous anticancer therapy, excluding hair changes such as alopecia or hair lightening.
* Currently pregnant (confirmed with positive pregnancy test) or breastfeeding (lactation must be discontinued throughout the period of the study and until at least one week after the last dose of study intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The number of treated patients with adverse events as determined by the common criteria for adverse version 5 (CTCAEv5). | 15 months
  We will be looking at safety and dose recommendations using adverse event evaluation per dose level as determined by CTCAEv5 (Part A)
Tumor response by imaging using RECISTv1.1 | 28 months
  We will determine the clinical benefit of this combination by evaluating tumor response by imaging using RECISTv1.1 guidelines (Part B)

SECONDARY OUTCOMES:
Percent apoptosis and tumor proliferation | 12 months
  To evaluate the percent apoptosis and tumor proliferation in resected tumor tissue ANNUBP after exposure to selumetinib and APG-115 (Part C)

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States